CLINICAL TRIAL: NCT00002132
Title: Randomized, Controlled, Double-Blind Study of Itraconazole Oral Solution Versus Fluconazole Tablets for the Treatment of Esophageal Candidiasis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 236A; ITR-USA-12
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Candidiasis, Esophageal; HIV Infections
Keywords: Itraconazole; Fluconazole; Acquired Immunodeficiency Syndrome; Candidiasis; Immunocompromised Host
MeSH Terms: conditions — Candidiasis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Itraconazole; Fluconazole

INTERVENTIONS:
Drug: Itraconazole
Drug: Fluconazole

SUMMARY:
To evaluate the safety and efficacy of itraconazole oral solution versus fluconazole tablets for the treatment of esophageal candidiasis in immunocompromised patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Esophageal candidiasis.
* Histological evidence of Candida spp. at baseline with confirmation by positive mycological culture.
* HIV infection or other predisposing risk factor.
* Life expectancy of at least 2 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancies of the head or neck, if the treatment or disease will interfere with response assessment.
* Evidence of systemic fungal infection.
* Underlying clinical condition that would preclude study completion.
* Judged to be unreliable in regard to following physician's directives.

Concurrent Medication:

Excluded:

* Rifampin.
* Rifabutin.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* Terfenadine.
* Astemizole.
* H2 blockers.
* Continual antacids.
* Any investigational drug (expanded access drugs are allowed).

Patients with the following prior conditions are excluded:

* History of significant hepatic abnormalities or clinical evidence of hepatic disease within 2 months prior to study entry.
* History of hypersensitivity to imidazole or azole compounds.

Prior Medication:

Excluded:

* Other orally administered antifungal therapy within 3 days prior to study entry.
* Any investigational drug within 1 month prior to study entry (expanded access drugs are allowed).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Dr Eskild A Petersen, Tucson, Arizona
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCSD Med Ctr, San Diego, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Wayne State Univ / Harper Hosp, Detroit, Michigan
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Infectious Diseases Association / Research Med Ctr, Kansas City, Missouri
  - Erie County Med Ctr, Buffalo, New York
  - Dr Douglas Dieterich, New York, New York
  - Montefiore Med Ctr, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Bowman Gray School of Medicine, Winston-Salem, North Carolina
  - Univ Hosps of Cleveland, Cleveland, Ohio
  - Austin Infectious Disease Consultants, Austin, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas

REFERENCES:
- [Background] Barbaro G, Barbarini G, Di Lorenzo G. Fluconazole compared with itraconazole in the treatment of esophageal candidiasis in AIDS patients: a double-blind, randomized, controlled clinical study. Scand J Infect Dis. 1995;27(6):613-7. doi: 10.3109/00365549509047076. PMID 8685642